CLINICAL TRIAL: NCT02215083
Title: L-glutamine Supplementation to Alleviate Symptoms of Taxane-Induced Neuropathy in Patients With Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient Patient Population
Sponsor: Eastern Regional Medical Center (Other)
Collaborators: TSPC America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERMC 13-32
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Neuropathy
Keywords: peripheral neuropathy; breast cancer; taxane induced peripheral neuropathy; chemotherapy induced peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-Glutamine (Experimental): All patients will receive 20-30 grams of l-glutamine daily for 9 weeks (+/- 1 week)
  Interventions: Dietary Supplement: L-glutamine

INTERVENTIONS:
Dietary Supplement: L-glutamine — 10,000mg by mouth, twice daily for nine weeks (± 7 days) with one permitted dose escalation to a maximum of 10,000mg by mouth three times daily.
  Other Names: Glutamine

SUMMARY:
The purpose of the study is to determine whether daily, high-dose administration of l-glutamine can reduce numbness and tingling caused by a taxane chemotherapy in patients with breast cancer.

DETAILED DESCRIPTION:
L-glutamine has previously been shown to help reduce the incidence of numbness and tingling in patients with breast cancer who are receiving taxane chemotherapies. However, no study to date looks at the effect of l-glutamine given after this numbness and tingling (called 'perihperhal neuropathy') has already occurred. We hypothesize that administration of this amino acid in l-glutamine naïve patients will result in a measureable reduction of their taxane-induced neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the breast
* Received at least one prior taxane-containing chemotherapy regimen which resulted in persistent taxane-induced peripheral neuropathy
* Anticipated survival of at least 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) = 0, 1, or 2
* The patient must have screening laboratory: Transaminases<2.5 x upper limit of normal; total bilirubin <2.0; creatinine <1.5
* Neuropathy onset from taxane administration no more than 18 months from date enrolled in trial
* Willingness to adhere to supplemental regimen of l-glutamine 10,000mg taken orally twice daily, with one potential dose escalation to 10,000mg taken orally three times daily.
* Grade I-III sensory peripheral neuropathy related to prior taxane use as assessed by their treating oncologist at Eastern Regional Medical Center
* Able to give informed consent for protocol participation

Exclusion Criteria:

* Participants are not able to understand or provide written informed consent.
* The research team deems that the participant may not be able to follow the study protocol.
* Current diagnosis of bipolar disorder or other manic state
* Prior use of l-glutamine for prevention or empirical treatment of taxane-induced sensory peripheral neuropathy
* Prior treatment with a platinum chemotherapy
* Concurrent use of physical therapy interventions such as the 'Rebuilder', chiropractic care, acupuncture, or other modalities specifically targeting peripheral neuropathy
* Concomitant use of nutraceutical supplements which may mitigate symptoms of taxane-induced peripheral neuropathy including B-Complex vitamins, alpha-lipoic acid, vitamin E, acetyl-l-carnitine, intramuscular B12 injections, fish oil, etc… during study
* Renal insufficiency : serum creatinine of >1.5 mg /dl
* Hepatic insufficiency: transaminases > 2.5 x upper limit of normal due to isolated reports of possible hepatic encephalopathy
* New prescription or dose adjustment of current medication for the treatment of peripheral neuropathy such as gabapentin or Lyrica within the past 30 days.
* Pre-existing sensory peripheral neuropathy from other comorbid conditions such as diabetes or alcoholism
* Current serious infection or other serious medical condition
* Currently active second malignancy other than nonmelanatous skin cancer or carcinoma in situ of the cervix
* Pregnant or lactating female (pre-menopausal females will undergo pregnancy test prior to administration of protocol drugs throughout treatment cycles during this study)
* Acetaminophen use exceeding 2 g per day-includes use of acetaminophen-containing pain medications such as Percocet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Total sensory neuropathy (area under the curve [AUC]) as measured by the EORTC QLQ-CIPN20 at baseline and week 9 | nine weeks

SECONDARY OUTCOMES:
Assess Quality of Life | nine weeks
  * Motor neuropathy as measured by the EORTC QLQ-CIPN20 at baseline and week 9
  * Autonomic symptoms and functioning as measured by the EORTC QLQ-CIPN20 at baseline and week 9
  * Overall quality of life as measured by the EORTC-30 questionnaire at baseline, 3 weeks, 6 weeks, and week 9
  * Pain severity as measured by the Visual Analog Numeric Pain Scale at baseline, week 3, week 6 and week 9
  * Objective assessment performed by Physical Therapy Department as measured by the Functional Gait Assessment at baseline and week 9
  * Frequency and severity of adverse events reported by the patient in the Symptom Experience Diary and evaluated through clinical assessment by NCI CTCAE v3.0

OTHER OUTCOMES:
Observe progression-free survival for 36 months post-intervention with l-glutamine supplementation | 40 months
  Quarterly record review to determine progression-free survival for 36 months post-l-glutamine intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jack Medendorp, Study Director — Eastern Regional Medical Center
Locations (1):
- Eastern Regional Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Stubblefield MD, Vahdat LT, Balmaceda CM, Troxel AB, Hesdorffer CS, Gooch CL. Glutamine as a neuroprotective agent in high-dose paclitaxel-induced peripheral neuropathy: a clinical and electrophysiologic study. Clin Oncol (R Coll Radiol). 2005 Jun;17(4):271-6. doi: 10.1016/j.clon.2004.11.014. PMID 15997923
- [Background] Vahdat L, Papadopoulos K, Lange D, Leuin S, Kaufman E, Donovan D, Frederick D, Bagiella E, Tiersten A, Nichols G, Garrett T, Savage D, Antman K, Hesdorffer CS, Balmaceda C. Reduction of paclitaxel-induced peripheral neuropathy with glutamine. Clin Cancer Res. 2001 May;7(5):1192-7. PMID 11350883